CLINICAL TRIAL: NCT03423355
Title: Dapagliflozin Effect on Erythropoiesis and Physical Fitness in Patients With Type 2 Diabetes - a Randomized, Partly Double-blinded, Controlled, Three Armed, Parallel Group, Exploratory Study
Brief Title: Dapagliflozin Effect on Erythropoiesis and Physical Fitness
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: change in sponsor
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DapaFIT
Record Dates: First submitted 2017-12-18; First posted 2018-02-06 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: Single center, prospective, randomized, double-blind, controlled, three-armed, parallel group, open-label reference group exploratory study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dapagliflozin (Forxiga®) (Active Comparator): Treatment with the SGLT2 inhibitor dapagliflozin 10 mg once daily for 28 days.
  Interventions: Drug: Dapagliflozin (Forxiga®)
- Placebo matching Dapagliflozin (Placebo Comparator): Treatment with the Dapagliflozin matching placebo once daily for 28 days.
  Interventions: Drug: Placebo matching Dapagliflozin
- Hydrochlorothiazide (Other): Treatment with the Hydrochlorothiazide 25 mg once daily for 28 days
  Interventions: Drug: Hydrochlorothiazide 25 mg

INTERVENTIONS:
Drug: Dapagliflozin (Forxiga®) — 10mg p.o. daily
  Arms: Dapagliflozin (Forxiga®)
Drug: Hydrochlorothiazide 25 mg — 25mg p.o. daily
  Arms: Hydrochlorothiazide
Drug: Placebo matching Dapagliflozin — Placebo matching Dapagliflozin p.o. daily
  Arms: Placebo matching Dapagliflozin

SUMMARY:
Dapagliflozin effect on erythropoiesis and physical fitness in patients with type 2 diabetes - a randomized, partly double-blinded, controlled, three armed, parallel group, exploratory study

DETAILED DESCRIPTION:
Many patients with diabetes present with hyperglycemia, hypertension, hypercholesterolemia and excess weight, which are associated with micro- and macrovascular complications. Therapies to alleviate the burden of these complications have traditionally focused on reducing glycemia and optimizing blood pressure and cholesterol concentration. However, despite the various available treatment options to improve glycemic control, many patients do not reach treatment and lifestyle targets, such as improving physical fitness. Sodium-glucose cotransporter 2 (SGLT2) inhibitors reduce the proximal tubule reabsorption of filtered glucose, thereby causing glucosuria and decreasing plasma glucose concentrations. When large quantities of glucose are pharmacologically forced into urinary excretion, whole-body metabolism undergoes adaptive changes, involving glucose fluxes, hormonal responses, fuel selection, and energy expenditure. SGLT2 inhibitors have been proven to be superior to conventional therapy by reducing cardiovascular mortality in patients with cardiovascular diseases (CVD). Many of the explained mechanisms contribute to this effect, and other, still unknown factors, need to be identified.

In the present study, patients suffering from T2DM and hypertension will be treated with Dapagliflozin, an SGLT2 inhibitor, or matching Placebo, or HCT as reference drug with a diuretic and anti-hypertensive effect.

There is evidence that SGLT2 inhibition positively affects the erythropoietin-RBC axis. By this mechanism, Dapagliflozin improves oxygen supply to tissues, an effect which can explain the positive cardiovascular (CV) outcome data of Dapagliflozin in recent registry data. The aim of the present study is to provide clinical endpoints related to this effect. Specifically, the effect of Dapagliflozin on erythropoietin, reticulocytes, and HIF related factors will be studied and related to physical fitness before and after treatment with Dapagliflozin. Providing evidence for an improvement in physical fitness and cardiac function by Dapagliflozin will be of great clinical benefit in patients with T2DM, since a large number of these patients have reduced physical activity and heart failure. The increasing effect of SGLT2 inhibitors on hematocrit was initially attributed to a relative hemoconcentration due to the diuretic effect elicited by the drug. However, studies comparing Dapagliflozin directly to diuretic treatment with HCT showed that the effect of Dapagliflozin was superior to diuretic treatment with HCT. Moreover, Dapagliflozin, and not HCT, also increased reticulocytes count and EPO concentrations [1]. Together, these data suggest that hemoconcentration is not mediating the effect of Dapagliflozin on hemopoiesis and that other mechanisms must contribute. Yet, reducing preload by diuretic properties may beneficially affect physical performance and may, thus, affect the secondary endpoint. Therefore, three treatments will be used in this study: Dapagliflozin and matching placebo, and HCT as reference treatment for the diuretic effect.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 40 and 70 years (including)
* Diagnosis of type 2 diabetes mellitus (T2DM) with HbA1c between 7.1 10.0% (including)
* Stable treatment of type 2 diabetes, except with SGLT2-Inhibitors over the last 4 weeks
* Body mass index (BMI) between 25 kg/m2 and 35 kg/m2 (including)
* Blood pressure > 130/80 mmHg but 170/95 mmHg at maximum
* Ability to perform spiroergometry
* Ability to understand and follow study-related instructions
* Negative pregnancy test
* Patients who are receiving the following medications must be on a stable treatment regimen for at least 2 months prior to the screening visit (V0): antihypertensive agents, thyroid replacement therapy, antidepressant agents

Exclusion Criteria:

* Diagnosis of Type 1 diabetes
* History of diabetic ketoacidosis, hyperosmolar coma or corticosteroid-induced T2DM
* Repeated episodes of severe hypoglycaemia within the last 3 months prior to Screening
* Patients with significant thyroid disease
* Intention to change physical activity within the next 8 weeks
* Clinically significant cardiovascular disease (CVD) or procedure within 3 months prior to enrollment or expected to require coronary revascularization procedure
* Presence of history of severe congestive heart failure (NYHA III and IV), pace maker or aortic stenosis (AS) > II
* eGFR (as calculated by the MDRD equation) < 60 ml/min/1.73 m2
* Unstable or rapidly progressing renal disease or anuria
* Concomitant medication with loop diuretics
* Any previous exposure to dapagliflozin or any other SGLT2-Inhibitor, or HCT within last 3 months prior to Screening
* Triglyceride concentrations ≥ 700 mg/dL (≥ 7.98 mmol/L) at the Screening visit (V0)
* History or presence of inflammatory bowel disease or other severe gastrointestinal diseases, particularly those which may impact gastric emptying, such as gastroparesis or pyloric stenosis
* History of gastric bypass surgery or gastric banding surgery, or either procedure is planned during the time period of the study. Current use of gastric balloons is also excluded
* • Significant hepatic disease, including, but not limited to, acute hepatitis, chronic active hepatitis, or severe hepatic insufficiency, including patients with alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3 x upper limit of normal (ULN) and/or total bilirubin (TB) > 2 mg/dL (> 34.2 μmol/L) (patients with TB > 2 mg/dL [> 34.2 μmol/L] and documented Gilbert's syndrome will be allowed to participate)
* Known human immunodeficiency virus (HIV) infection
* History of organ transplantation
* Malignancy (with the exception of basal and squamous cell carcinoma of the skin) within 5 years prior to the Screening visit (V1)
* • Hemoglobinopathy, hemolytic anemia, or chronic anemia (hemoglobin concentration < 12.0 g/dL) or any other condition known to interfere with the HbA1c methodology
* Patients who have donated blood or had a significant blood loss within 2 months of first dose of study medication or is planning to donate blood during the study
* Patients who have donated plasma within 7 days prior to first dose of study medication
* Systemic corticosteroids within 3 months prior to the Screening visit (V0) known to have a high rate of systemic absorption
* History of chronic obstructive pulmonary disease (COPD) or asthma
* Disabilities contraindicating spiroergometry
* Alcohol consumption > 20 g/day for women or > 30 g/day for men
* History of hypersensitivity to any of the study drugs or their ingredients
* Presence of psychiatric disorder or intake of anti-depressive or anti-psychotic agents with the exception of benzodiazepines and SSRIs/SNRI´s
* Addiction or other diseases that preclude the patient from appropriately assessing the nature and scope as well as possible consequences of the clinical study
* Pregnant or breastfeeding women
* Subject (male or female) is not willing to use highly effective contraceptive methods during treatment and for 14 days (male or female) after the end of treatment (highly effective methods are defined as: combined hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence). Vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the trial participant and that the vasectomized partner has received medical assessment of the surgical success In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
* Participation in other clinical trials

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood EPO levels | 2 weeks of treatment
  The primary objective is to investigate the change in erythropoietin (EPO) levels after 2 weeks of treatment with dapagliflozin in comparison to treatment with placebo.

SECONDARY OUTCOMES:
Change in physical fitness | 4 weeks of treatment
  Change in physical fitness between baseline and EoT as assessed by spiroergometry (VO2max, heart rate and blood pressure) with dapagliflozin in comparison to treatment with placebo
Change in reticulocyte concentration, hematocrit and red blood cells | baseline, 2 weeks and 4 weeks of treatment
  Change in reticulocyte concentration, hematocrit and red blood cells between baseline and after 2 and 4 weeks of treatment with dapagliflozin in comparison to treatment with placebo
Change in hepcidin | baseline and 4 weeks of treatment
  Change in hepcidin between baseline and EoT with dapagliflozin in comparison to treatment with placebo
Change in blood EPO levels | baseline, 4 weeks of treatment
  Change in blood EPO levels between baseline and EoT (comparison dapagliflozin vs HCT vs placebo)
Change in iron status (Fe) | baseline and 4 weeks of treatment
  Change in iron status between baseline and EoT as measured by Fe with dapagliflozin in comparison to treatment with placebo
Change in iron status (Ferritin) | baseline and 4 weeks of treatment
  Change in iron status between baseline and EoT as measured by ferritin with dapagliflozin in comparison to treatment with placebo
Change in iron status (Transferrin) | baseline and 4 weeks of treatment
  Change in iron status between baseline and EoT as measured by transferrin with dapagliflozin in comparison to treatment with placebo
Change in catecholamine (adrenalin) | baseline and 4 weeks of treatment
  Change in adrenalin concentrations between baseline and EoT with dapagliflozin in comparison to treatment with placebo
Change in catecholamine (noradrenalin) | baseline and 4 weeks of treatment
  Change in noradrenalin concentrations between baseline and EoT with dapagliflozin in comparison to treatment with placebo
Change in catecholamine (metabolites metanephrine) | baseline and 4 weeks of treatment
  Change in metabolites metanephrine concentrations between baseline and EoT with dapagliflozin in comparison to treatment with placebo
Change in catecholamine (normetanephrine) | baseline and 4 weeks of treatment
  Change in normetanephrine concentrations between baseline and EoT with dapagliflozin in comparison to treatment with placebo
Change in steroid hormone | baseline and 4 weeks of treatment
  Change in steroid hormone concentrations between baseline and EoT with dapagliflozin in comparison to treatment with placebo
Change of ejection fraction | baseline and 4 weeks of treatment
  Change of ejection fraction measured by echocardiography, between baseline and EoT with dapagliflozin in comparison to treatment with placebo
Change of diastolic function parameters | baseline and 4 weeks of treatment
  Change of diastolic function parameters measured by echocardiography, between baseline and EoT with dapagliflozin in comparison to treatment with placebo

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Otfried-Mueller Str. 10, Tübingen, Germany